CLINICAL TRIAL: NCT02218580
Title: Massage Therapy for Children With Juvenile Idiopathic Arthritis Experiencing Pain: a Pilot Randomized Controlled Trial
Brief Title: Massage Therapy in Juvenile Idiopathic Arthritis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit study participants
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Sarah Campillo, Pediatric Rheumatologist, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRA (CIORA grant #4)
Record Dates: First submitted 2014-07-07; First posted 2014-08-18 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: massage therapy; juvenile arthritis; pain
MeSH Terms: conditions — Arthritis, Juvenile; Pain | interventions — Massage; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Massage therapy & standard care (Experimental): Massage therapy will be provided by caregiver for 15 minutes at bedtime at home, every night, for a 2-week period.
  Standard care will include medications routinely prescribed in the treatment of JIA, physiotherapy and occupational therapy exercises, splints, warmth application and acetaminophen.
  Interventions: Other: Massage therapy; Other: Standard care
- Standard care (Active Comparator): Standard care will include medications routinely prescribed in the treatment of JIA, physiotherapy and occupational therapy exercises, splints, warmth application and acetaminophen.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Massage therapy
  Arms: Massage therapy & standard care
Other: Standard care

SUMMARY:
While there has been progress in juvenile idiopathic arthritis (JIA) management, there is no cure. Despite receiving standard of care, many children live with pain. Thus, it is not surprising that families turn to complementary and alternative medicines (CAM) therapies, including massage therapy (MT). Little is known about the efficacy of MT in JIA.

In this project, a massage therapist will teach parents how to provide a massage to their child with JIA at bedtime, at home. The feasibility of establishing a home MT program for children with JIA will be evaluated. In addition, the effects of MT on JIA will be examined.

This proposal is relevant to JIA families, who ask questions on MT to professionals of the JIA clinic.

Beyond providing education to JIA families, this project demonstrates the team approach to JIA management. Team members will include a pediatric rheumatology nurse and a massage therapist.

DETAILED DESCRIPTION:
While research breakthroughs have led to improved outcomes, many patients with JIA live with pain. There is an association between daily fluctuations in JIA symptoms (pain, stiffness and fatigue), and worse mood and stressful events, supporting the utility of daily diaries to analyze JIA symptoms. Sleep disturbances have been demonstrated in JIA and are linked to the pain experience. Ultimately, pain impacts on HRQoL. JIA families explore complementary and alternative medicines such as MT, in addition to using conventional medicines, to help manage the daily JIA symptoms. MT's effects on pain, mood, anxiety, stress and sleep have been demonstrated in several diseases, possibly through modulation of neurological, endocrine and immune processes. Children with JIA and pain could benefit from MT given with standard care. Only one study evaluated its benefits in JIA. More research is needed on the feasibility, efficacy and safety of MT in JIA. MT is available at the Montreal Children's Hospital in Oncology. While offering MT in the hospital setting is practical for oncology patients who require frequent hospitalizations, MT may be more beneficial for JIA patients if implemented at home.

Objectives The primary purpose of this single center, pilot randomized controlled trial (pilot RCT) is to determine the feasibility of a home MT program for children with JIA experiencing pain. The second purpose is to determine the effects of MT primarily on daily pain, as well as, other daily JIA symptoms (stiffness and fatigue), sleep quality, health-related quality of life (HRQoL) and disease activity, and on caregiver's psychological distress. The effects of MT on pro-inflammatory cytokines (IL-6, 17A, TNF) will be explored.

Methodology During the pilot RCT (Part 1), 30 children with JIA who experience pain will be randomized to the experimental group (home MT and standard care) or control group (standard care). After receiving training by the massage therapist, caregivers of the experimental group will gently massage their child, for 15 minutes at bedtime, every night, at home. Immediately after the RCT, participants of the control group will receive training and implement home MT, similar to the experimental group, in an extension (Part 2).

Feasibility will be evaluated by the recruitment rate, retention rate, program adherence, piloting of the intervention, and user acceptability and satisfaction with the program.

Given the daily fluctuations in JIA symptoms, daily pain, fatigue, stiffness and sleep quality will be evaluated through multiple measurements with daily diaries to be completed by patients and their caregivers, both before and after implementation of home MT in both groups. Sleep, fatigue, HRQoL, disease activity and caregiver's psychological distress will also be evaluated before and after implementation of home MT in both groups, with questionnaires, physical examinations and blood samples.

Conclusion The findings from this project will provide the framework for planning a multi-center study whose focus will be on the efficacy of MT in JIA. MT programs do not exist in Canadian pediatric rheumatology centres and thus, this project is innovative. If there is preliminary evidence that MT helps reduce pain, it could become an additional strategy to help these children have a better HRQoL, with less pain and improved health outcomes. Parents could feel empowered by participating concretely and in a positive way in the management of their child's condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of JIA (ILAR classification)
* Age 5 to 17 years
* Ability to speak/read French or English; one caregiver per child will be recruited;
* Presence of pain, defined as: pain reported by the child and/or caregiver, and/or joint tenderness and/or stress pain in at least 1 joint during physical examination performed by rheumatologist. Pain reported by the child/caregiver is not a prerequisite because some children develop behaviors and guarding postures to avoid pain
* Absence of anticipated change in treatment. If, during the study, a change in treatment is necessary, the change will be recorded but the child will not be withdrawn
* Stable dosages of medications and absence of intra-articular corticosteroid injections for 4 weeks prior to enrolment
* Eligibility confirmed by child's rheumatologist.

Exclusion Criteria:

* No current MT
* Systemic arthritis with quotidian fevers
* Acute infection
* Open skin lesion
* Fibromyalgia
* Sleep apnea
* Medications: anticoagulants, muscle relaxants, analgesic medications (acetaminophen allowed)
* Pregnancy.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2015-05; Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 1 year
  Recruitment rate will be measured to evaluate the feasibility of a home MT program. The recruitment rate is defined as the proportion of patients recruited out of eligible patients.
Retention rate | 1 year
  Retention rate will be measured to evaluate the feasibility of a home MT program. Retention rate is defined as the proportion of patients who complete the MT program.
Program adherence | 1 year
  Program adherence will be measured to evaluate the feasibility of a home MT program. Program adherence is defined as the proportion of daily diaries completed by families.
Piloting the intervention | 1 year
  Suggestions for program improvement from massage therapist, research coordinator, nurse and investigators will be recorded, in order to evaluate the feasibility of a home MT program.
User acceptability and satisfaction | 1 year
  User acceptability and satisfaction will be evaluated to assess the feasibility of a home MT program. Caregivers will be asked to evaluate the helpfulness and ease of implementation of the program, provide suggestions for improvement, indicate whether they would recommend it to others.

SECONDARY OUTCOMES:
Daily pain | Daily for 4 weeks for the intervention group and for 6 weeks for the control group
  Daily pain will be measured on 100 mm visual analogue scales (VAS) with the use of daily diaries, completed on a daily basis. Daily pain will be assessed in the evening. Caregivers and children over 8 years will complete VAS. All children will also complete the Faces Pain Scaled-Revised and will record painful locations on a body map. In the intervention group, the diaries will be completed every day, for a 2 week period before implementation of massage therapy, and for a 2 week period following implementation of massage therapy. In the control group, the diaries will be completed every day, for a 4 week period before implementation of massage therapy, and for a 2 week period following implementation of massage therapy.
Daily fatigue | Daily for 4 weeks for the intervention group and for 6 weeks for the control group
  Daily fatigue will be measured on 100 mm VAS with the use of daily diaries, completed on a daily basis. Fatigue will be assessed in the evening. Caregivers and children over 8 years will complete VAS. In the intervention group, the diaries will be completed every day, for a 2 week period before implementation of massage therapy, and for a 2 week period following implementation of massage therapy. In the control group, the diaries will be completed every day, for a 4 week period before implementation of massage therapy, and for a 2 week period following implementation of massage therapy.
Daily stiffness | Daily for 4 weeks for the intervention group and for 6 weeks for the control group
  Daily stiffness will be measured on 100mm VAS with the use of daily diaries, completed on a daily basis. Stiffness will be assessed in the evening. Caregivers and children over 8 years will complete VAS. In the intervention group, the diaries will be completed every day, for a 2 week period before implementation of massage therapy, and for a 2 week period following implementation of massage therapy. In the control group, the diaries will be completed every day, for a 4 week period before implementation of massage therapy, and for a 2 week period following implementation of massage therapy.
Daily sleep quality | Daily for 4 weeks for the intervention group and for 6 weeks for the control group
  Daily sleep quality will be measured on 100mm VAS with the use of daily diaries, completed on a daily basis. Daily sleep quality will be assessed in the morning. Caregivers and children over 8 years will complete VAS. In the intervention group, the diaries will be completed every day, for a 2 week period before implementation of massage therapy, and for a 2 week period following implementation of massage therapy. In the control group, the diaries will be completed every day, for a 4 week period before implementation of massage therapy, and for a 2 week period following implementation of massage therapy.
Health-related Quality of Life (HRQOL) | HRQOL will be measured three times during a 4 week period for the intervention group (Day 1, Day 15 and Day 29) and a 6 week period for the control group (Day 1, Day 30 and Day 44).
  HRQOL will be measured by questionnaires, using the Pediatric Quality of Life Inventory (PedsQL) 4.0 Generic Core Scales and the PedsQL 3.0 Rheumatology module. Both caregivers and children will complete the questionnaires, at 3 time points (before implementation of MT, on the MT training day and after implementation of MT).
Fatigue | Fatigue will be measured three times during a 4 week period for the intervention group (Day 1, Day 15 and Day 29) and a 6 week period for the control group (Day 1, Day 30 and Day 44).
  Fatigue will be measured by a questionnaire, using the PedsQL Multidimensional Fatigue Scale. Both caregivers and children will complete the questionnaire, at 3 time points (before implementation of MT, on the MT training day and after implementation of MT).
Sleep quality | Sleep quality will be measured three times during a 4 week period for the intervention group (Day 1, Day 15 and Day 29) and a 6 week period for the control group (Day 1, Day 30 and Day 44).
  Sleep quality will be measured by a questionnaire, using the Sleep Disturbance Scale for Children. Caregivers will complete this questionnaire, at 3 time points (before implementation of MT, on the MT training day and after implementation of MT).
Caregiver's psychological distress | Caregiver's psychological distress will be measured three times during a 4 week period for the intervention group (Day 1, Day 15 and Day 29) and a 6 week period for the control group (Day 1, Day 30 and Day 44).
  Caregiver's psychological distress will be measured by a questionnaire, using the Symptom Checklist-90-Revised. Caregivers will complete this questionnaire, at 3 time points (before implementation of MT, on the MT training day and after implementation of MT).
Disease activity | Disease activity will be evaluated before and after implementation of MT: on Day 1 and Day 29 for the intervention group; and on Day 1 and Day 44 for the control group.
  Disease activity will be evaluated with the active joint count (AJC) and the physician global assessment of disease activity (PGADA), obtained by physical examination performed by the rheumatologist. Disease activity will also be evaluated by the erythrocyte sedimentation rate (ESR) and the C-reactive protein (CRP), obtained by blood tests.

OTHER OUTCOMES:
Levels of pro-inflammatory cytokines (IL-6, IL-17a, TNF) | Levels of pro-inflammatory cytokines will be evaluated before and after implementation of MT: on Day 1 and Day 29 for the intervention group; and on Day 1 and Day 44 for the control group.
  The effects of MT on pro-inflammatory cytokines (IL-6, IL-17a, TNF) will be explored. Cytokines produced by stimulated cells isolated from whole blood will be measured by BD Cytometric Bead Array.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Campillo, MD, Principal Investigator — Montreal Children's Hospital of the MUHC
Locations (1):
- Montreal Children's Hospital - Glen site, Montreal, Quebec, Canada

REFERENCES:
- [Background] Bromberg MH, Connelly M, Anthony KK, Gil KM, Schanberg LE. Self-reported pain and disease symptoms persist in juvenile idiopathic arthritis despite treatment advances: an electronic diary study. Arthritis Rheumatol. 2014 Feb;66(2):462-9. doi: 10.1002/art.38223. PMID 24504820
- [Background] Schanberg LE, Anthony KK, Gil KM, Maurin EC. Daily pain and symptoms in children with polyarticular arthritis. Arthritis Rheum. 2003 May;48(5):1390-7. doi: 10.1002/art.10986. PMID 12746912
- [Background] Schanberg LE, Gil KM, Anthony KK, Yow E, Rochon J. Pain, stiffness, and fatigue in juvenile polyarticular arthritis: contemporaneous stressful events and mood as predictors. Arthritis Rheum. 2005 Apr;52(4):1196-204. doi: 10.1002/art.20952. PMID 15818661
- [Background] Bloom BJ, Owens JA, McGuinn M, Nobile C, Schaeffer L, Alario AJ. Sleep and its relationship to pain, dysfunction, and disease activity in juvenile rheumatoid arthritis. J Rheumatol. 2002 Jan;29(1):169-73. PMID 11824956
- [Background] Passarelli CM, Roizenblatt S, Len CA, Moreira GA, Lopes MC, Guilleminault C, Tufik S, Hilario MO. A case-control sleep study in children with polyarticular juvenile rheumatoid arthritis. J Rheumatol. 2006 Apr;33(4):796-802. Epub 2006 Mar 1. PMID 16511937
- [Background] Oliveira S, Ravelli A, Pistorio A, Castell E, Malattia C, Prieur AM, Saad-Magalhaes C, Murray KJ, Bae SC, Joos R, Foeldvari I, Duarte-Salazar C, Wulffraat N, Lahdenne P, Dolezalova P, de Inocencio J, Kanakoudi-Tsakalidou F, Hofer M, Nikishina I, Ozdogan H, Hashkes PJ, Landgraf JM, Martini A, Ruperto N; Pediatric Rheumatology International Trials Organization (PRINTO). Proxy-reported health-related quality of life of patients with juvenile idiopathic arthritis: the Pediatric Rheumatology International Trials Organization multinational quality of life cohort study. Arthritis Rheum. 2007 Feb 15;57(1):35-43. doi: 10.1002/art.22473. PMID 17266064
- [Background] Shaw KL, Southwood TR, McDonagh JE. Growing up and moving on in rheumatology: parents as proxies of adolescents with juvenile idiopathic arthritis. Arthritis Rheum. 2006 Apr 15;55(2):189-98. doi: 10.1002/art.21834. PMID 16583398
- [Background] April KT, Feldman DE, Zunzunegui MV, Descarreaux M, Malleson P, Duffy CM. Longitudinal analysis of complementary and alternative health care use in children with juvenile idiopathic arthritis. Complement Ther Med. 2009 Aug;17(4):208-15. doi: 10.1016/j.ctim.2009.03.003. Epub 2009 May 1. PMID 19632548
- [Background] van Tulder MW, Furlan AD, Gagnier JJ. Complementary and alternative therapies for low back pain. Best Pract Res Clin Rheumatol. 2005 Aug;19(4):639-54. doi: 10.1016/j.berh.2005.03.006. PMID 15949781
- [Background] Kalichman L. Massage therapy for fibromyalgia symptoms. Rheumatol Int. 2010 Jul;30(9):1151-7. doi: 10.1007/s00296-010-1409-2. Epub 2010 Mar 20. PMID 20306046
- [Background] Bender T, Nagy G, Barna I, Tefner I, Kadas E, Geher P. The effect of physical therapy on beta-endorphin levels. Eur J Appl Physiol. 2007 Jul;100(4):371-82. doi: 10.1007/s00421-007-0469-9. Epub 2007 May 5. PMID 17483960
- [Background] Sunshine W, Field TM, Quintino O, Fierro K, Kuhn C, Burman I, Schanberg S. Fibromyalgia benefits from massage therapy and transcutaneous electrical stimulation. J Clin Rheumatol. 1996 Feb;2(1):18-22. doi: 10.1097/00124743-199602000-00005. PMID 19078022
- [Background] Diego MA, Field T, Hernandez-Reif M, Shaw K, Friedman L, Ironson G. HIV adolescents show improved immune function following massage therapy. Int J Neurosci. 2001 Jan;106(1-2):35-45. doi: 10.3109/00207450109149736. PMID 11264907
- [Background] Field T, Morrow C, Valdeon C, Larson S, Kuhn C, Schanberg S. Massage reduces anxiety in child and adolescent psychiatric patients. J Am Acad Child Adolesc Psychiatry. 1992 Jan;31(1):125-31. doi: 10.1097/00004583-199201000-00019. PMID 1537763
- [Background] Field T, Henteleff T, Hernandez-Reif M, Martinez E, Mavunda K, Kuhn C, Schanberg S. Children with asthma have improved pulmonary functions after massage therapy. J Pediatr. 1998 May;132(5):854-8. doi: 10.1016/s0022-3476(98)70317-8. PMID 9602199
- [Background] Hart S, Field T, Hernandez-Reif M, Nearing G, Shaw S, Schanberg S, Kuhn C. Anorexia nervosa symptoms are reduced by massage therapy. Eat Disord. 2001 Winter;9(4):289-99. doi: 10.1080/106402601753454868. PMID 16864390
- [Background] Field T, Hernandez-Reif M, Seligman S, Krasnegor J, Sunshine W, Rivas-Chacon R, Schanberg S, Kuhn C. Juvenile rheumatoid arthritis: benefits from massage therapy. J Pediatr Psychol. 1997 Oct;22(5):607-17. doi: 10.1093/jpepsy/22.5.607. PMID 9383925
- [Background] Field T. Massage therapy for infants and children. J Dev Behav Pediatr. 1995 Apr;16(2):105-11. PMID 7790516